CLINICAL TRIAL: NCT01236378
Title: An Open-Label, Non-Randomized Study To Evaluate The Steady-State Pharmacokinetics Of Sirolimus Tablets In Chinese Patients With Stable Renal Allografts
Brief Title: Study To Evaluate Pharmacokinetics Of Sirolimus In Stable Renal Transplant Recipients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1741018
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2011-04

CONDITIONS: Transplant Rejection; Renal Transplantation
Keywords: Organ Transplants; Anti-Rejection Therapy; Pharmacokinetics
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sirolimus (Experimental): Subjects must be taking sirolimus (1 mg tablet formulation) with or without concomitant medications, unless specifically excluded below, for prophylaxis of renal rejection.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus, 1 mg, white, triangular tablets, daily dose, dosages of any of these medications must be stable for at least 2 weeks prior to screening and continue with no change until completion of the last PK sample collection.
  Other Names: Rapamune

SUMMARY:
Sirolimus, 1 mg, white, triangular tablets (Rapamune®) was approved on 03 April 2007 in China for prophylaxis of organ rejection in renal transplantation. A pharmacokinetic (PK) study to be conducted in renal allograft recipients was requested by State Food and Drug Administration (SFDA) to provide further guidance for clinical use.

To minimize risk to patients, this study is designed to collect blood PK samples from renal allograft recipients who are currently under sirolimus (1 mg tablets) treatment with or without concomitant medication(s). PK samples will be collected from these patients to characterize the steady state PK of sirolimus during sirolimus maintenance therapy. This study will not involve any changes to the established treatment regimen for the patients who enroll in the study

ELIGIBILITY:
Inclusion Criteria:

* Male or female, above 18 years of age and Body Mass Index (BMI) of 18.0 to 25.0 kg/m2, inclusive;
* Subjects must have received a primary or secondary renal allograft for at least 2 months prior to Screening;
* Subjects must be currently taking Rapamune tablets for prophylaxis of renal rejection. The dosages of any medications must be stable for at least 2 weeks prior to screening and continue with no change until completion of the last PK sample collection.

Exclusion Criteria:

* Acute rejection or vascular rejection episode in the 4 weeks prior to Screening; or patients dependent on dialysis; or inadequate renal function (in the opinion of the investigator);
* Recipients of multiple organ transplants (i.e., prior or concurrent transplantation of any organs other than renal transplant);
* Current use of strong inducers or inhibitors of CYP3A4 within 2 weeks prior to collection of the first PK sample and until collection of the final PK sample;
* Any clinically significant medical or psychiatric condition or laboratory abnormality, in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Pfizer Investigational Site, Chongqing
  - Pfizer Investigational Site, Shanghai

REFERENCES:
- [Derived] Wang HF, Qiu F, Wu X, Fang J, Crownover P, Korth-Bradley J, Schulman S. Steady-state pharmacokinetics of sirolimus in stable adult Chinese renal transplant patients. Clin Pharmacol Drug Dev. 2014 May;3(3):235-41. doi: 10.1002/cpdd.96. Epub 2014 Feb 10. PMID 27128614
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1741018&StudyName=Study%20To%20Evaluate%20Pharmacokinetics%20Of%20Sirolimus%20In%20Stable%20Renal%20Transplant%20Recipients

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus: Sirolimus, 1 milligram (mg) tablet formulation; total daily dosage could have varied from participant to participant, dosage must have been stable for at least 2 weeks prior to screening and continued with no change until completion of the last pharmacokinetic (PK) sample collection.
Period: Overall Study
Arm/Group | Sirolimus
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sirolimus: Sirolimus, 1 mg tablet formulation; total daily dosage could have varied from participant to participant, dosage must have been stable for at least 2 weeks prior to screening and continued with no change until completion of the last PK sample collection.
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
Age, Customized [Number; unit: participants]
  18 to 44 years | 16
  45 to 64 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Blood Concentration at Steady State (Cmax,ss)
Time Frame: Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours post dose
Population: PK parameter analysis population: All treated participants who had at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
nanogram per milliliter (ng/mL) | 14.07 (13.433)

2. Primary Outcome: Time to Reach Maximum Observed Blood Concentration at Steady State (Tmax,ss)
Time Frame: Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours post dose
Population: PK Parameter Analysis Population
Measure: Median (Full Range); unit: hours
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
hours | 2.49 [0.983 to 12.0]

3. Primary Outcome: Observed Blood Trough Concentration at Steady State (Ctrough,ss)
Time Frame: Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours post dose
Population: PK Parameter Analysis Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
ng/mL | 5.906 (6.2621)

4. Primary Outcome: Average Blood Concentration at Steady State (Cave,ss)
Time Frame: Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours post dose
Population: PK Parameter Analysis Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
ng/mL | 8.297 (8.7384)

5. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) at Steady State
Time Frame: Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours post dose
Population: PK Parameter Analysis Population
Measure: Mean (Standard Deviation); unit: nanogram hour per milliliter (ng*h/mL)
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
nanogram hour per milliliter (ng*h/mL) | 199.3 (209.96)

6. Primary Outcome: Degree of Fluctuation (DF)
Description: DF, also known as peak to trough fluctuation (PTF) (calculated as [Cmax minus Ctrough] divided by Cave), is a unit-less ratio of the Cmax to Ctrough decrease expressed as a fraction of the average concentration during a dosing interval.
Time Frame: Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours post dose
Population: PK Parameter Analysis Population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
ratio | 1.064 (0.3226)

7. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours post dose
Population: PK Parameter Analysis Population
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
liter per hour (L/h) | 10.14 (4.3678)

8. Secondary Outcome: Number of Participants With Serum Creatinine Levels More Than (>) 1.3 Times the Upper Limit of Normal
Description: Serum creatinine, an indicator of kidney function, formed from the metabolism of creatine, commonly found in blood, urine, and muscle tissue, is removed from blood by kidneys and excreted in urine. Increased creatinine in blood indicates decreased kidney function. Creatinine levels are age, gender and race dependent as they are related to an individual's muscle mass. Renal transplant recipients may have elevated serum creatinine. For this study an abnormal serum creatinine level is defined as 1.3 times the upper limit of normal (ULN) for the laboratory where the determination was performed.
Time Frame: From baseline up to Day 4
Population: All participants.
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
participants
  Baseline | 5
  Day 4 | 4

9. Secondary Outcome: Number of Participants With Estimated Glomerular Filtration Rate (GFR) Less Than (<) 60 mL/Min/1.73 m^2
Description: GFR, an index of kidney function, describes flow rate of filtered fluid through the kidney. GFR can be measured directly or estimated using established formulas. GFR was calculated using the Simplified Modification of Diet in Renal Dysfunction (MDRD) GFR equation. Normal GFR is >90 mL/min/1.73 m^2; children and older people usually have lower GFR. Often, kidney transplant recipients do not have normal GFRs. Lower values indicate poor kidney function. GFR <15 mL/min/1.73 m^2 is consistent with kidney failure. For this posting, the number of subjects with a GFR <60 mL/min/1.73 m^2 is listed.
Time Frame: From baseline up to Day 4
Population: All participants.
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
participants
  Baseline | 7
  Day 4 | 7

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sirolimus
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.